CLINICAL TRIAL: NCT05773573
Title: Comparison of Skeletal and Dental Changes with Hyrax-type Rapid Maxillary Expander Anchored to Permanent (6) Versus Deciduous Molars (V) in Growing Subjects
Brief Title: Skeletal and Dental Changes with Hyrax-type Rapid Maxillary Expander Anchored to Permanent Versus Deciduous Molars
Acronym: DENTHYRAX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL22_0144
Record Dates: First submitted 2023-03-06; First posted 2023-03-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Maxillary Hypoplasia
Keywords: Orthodontic appliances; Orthodontic interceptive; Palatal expansion technique; Child; Dentition mixed; Tooth deciduous; Rapid maxillary expansion
MeSH Terms: conditions — Retrognathia | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Hyrax-type rapid maxillary expander anchored on the 2nd deciduous molars (V)
  Interventions: Device: Experimental group
- Control group (Active Comparator): Hyrax-type rapid maxillary expander anchored on the 1st permanent molars (6)
  Interventions: Device: Control group

INTERVENTIONS:
Device: Experimental group — The experimental group will have a hyrax rapid maxillary expander anchored on the 2nd deciduous molars (V)
  Arms: Experimental group
Device: Control group — The control group will have a hyrax rapid maxillary expander anchored on the 1st permanent molars (6)
  Arms: Control group

SUMMARY:
The aim of the study is to compare the skeletal and dental maxillary expansion obtained with an Hyrax tooth-borne expander anchored either on the 2nd deciduous molars (V) or on the 1st permanent molars (6)

DETAILED DESCRIPTION:
The aim of the study is to compare the skeletal and dental maxillary expansion obtained with an Hyrax tooth-borne expander anchored either on the 2nd deciduous molars (V) or on the 1st permanent molars (6).

The main objective is to compare at the skeletal level the distance between the cephalometric points, right jugal (RJ) and left jugal (JR) (maxillary base).

The secondaries objectives are performed at the dental level by measuring the distance between the maxillary first molars mesio-palatal cusp and the cuspids cups. Molar derotation is also assessed

ELIGIBILITY:
Inclusion Criteria:

* Patient coming to the dental clinic for a first orthodontic consultation in mixed dentition
* Patient aged 6 to 12 years
* Patient with a transverse maxillary deficiency requiring rapid maxillary expansion
* Presence of 1st permanent molars "6" and 2nd deciduous "V" molars with sufficient root length

Exclusion Criteria:

* Syndromic patients (all syndromes combined: cleft lip, etc.)
* Patient with V or 6 with decays (or with major root resorption)
* Patient with oral hygiene non compatible with orthodontic treatment
* Failure to obtain informed written consent
* No affiliation to a French national medical health system
* Patient with a legal protection measure

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Difference in skeletal maxillary width before/ after rapid maxillary expansion | 6 months
  Difference in skeletal maxillary width measured on frontal cephs (distance between the cephalometric points "right jugal RJ" and "left jugal JR" of the Ricketts analysis) before (V0)/after (V8) rapid maxillary expansion with tooth-borne expander type Hyrax

SECONDARY OUTCOMES:
Difference of the inter-molar distance before/after | 6 months
  Difference before (V0) / after (V8) rapid maxillary expansion with tooth-borne expander type Hyrax of the inter-molar distance (mesiopalatal cusp) assessed on dental casts
Difference of the inter-canine distance before/after | 6 months
  Difference before (V0) / after (V8) rapid maxillary expansion with tooth-borne expander type Hyrax of the inter-canine distance (cuspids cusp) assessed on dental casts
Difference in the amount of molar derotation (inter-molar angle) before/after | 6 months
  Difference before (V0) / after (V8) rapid maxillary expansion with tooth-borne expander type Hyrax in the amount of molar derotation (inter-molar angle) assessed on dental casts
Inter-operator reproducibility | 1 month
  Inter-operator reproducibility assessed by the intra-class correlation coefficient

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Soins Dentaires, Montpellier, France

IPD SHARING:
Plan to Share IPD: No